CLINICAL TRIAL: NCT00288158
Title: Primary Prevention of Hypertension in Obese Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK71223 (completed); R21DK071223 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Pre-Hypertension; Hyperuricemia
MeSH Terms: conditions — Obesity; Prehypertension; Hyperuricemia | interventions — Allopurinol; Probenecid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Allopurinol (Experimental)
  Interventions: Drug: Allopurinol
- Probenecid (Experimental)
  Interventions: Drug: Probenecid
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol
  Arms: Allopurinol
Drug: Probenecid
  Arms: Probenecid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the consequences of lowering serum uric acid in pre-hypertensive, obese adolescents pathways involved with how uric acid mediated hypertension and renal disease. The specific aims are:

1. Test the hypothesis that lowering uric acid will improve endothelial function.
2. Test the hypothesis that lowering uric acid will reduce plasma renin activity and serum angiotensin II levels.
3. Test the hypothesis that lowering uric acid will reduce markers of inflammation

DETAILED DESCRIPTION:
The trial will be a double blinded, placebo control trial of two uric acid lowering agents. The endpoints for this trial will be, endothelial function, systemic vascular resistance, plasma renin activity, MCP-1 and CRP. Upon recruitment and informed consent, children will undergo initial screening. This will include medical history, family history, dietary history, review of systems (questionnaire used and validated in pediatric hypertension clinic) and pediatric quality of life questionnaire. They will have a physical exam, casual and ambulatory blood pressure monitoring (see below) and screening laboratory analysis that will include CBC, electrolytes, BUN, Cr, Uric acid, AST, ALT and urinary micro-albumin to creatinine ratio. Children with serum uric acid less than 5.0mg per dl will be enrolled as controls and only have baseline studies at Screening and Visit 1. Children with serum uric acid equal to or greater than 5.0mg per dl will be randomized (in a one to one to one ratio) to receive placebo, allopurinol or probenecid.

Study drug (or placebo) will be administered for 2 months. During the first week, subjects will take one tablet (placebo, 150mg allopurinol or 250mg probenecid) twice daily. At the end of one week subjects will be instructed to increase to 2 tablets (placebo, 300mg allopurinol or 500mg probenecid) twice daily. Data collection will occur during screening, after one and two months on the study drug and one month after completion of the study drug.

ELIGIBILITY:
Inclusion Criteria:

Children between the ages of 11 and 18

body mass index greater than the 95th percentile for age

Blood pressure between 75th and 95th percentile for age, gender and height percentile

Exclusion Criteria:

hypertension at the time of screening

allergy to one of the study medications

liver function abnormality (AST or ALT greater than twice the upper limit of

normal for the laboratory)

history of renal stones

renal insufficiency (Schwartz formula calculated GFR less than 70ml per min per 1.73m2 BSA)

positive urine pregnancy test

diabetes

organ transplant recipient

currently treated with an angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), diuretic, other medications known to alter serum uric acid level

lack of ability to comply with the study protocol

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Casual BP | 3 months

SECONDARY OUTCOMES:
24- hour Ambulatory BP | 3 months
Systemic Vascular Resistance (measured by bioimpedance) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Feig, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Soletsky B, Feig DI. Uric acid reduction rectifies prehypertension in obese adolescents. Hypertension. 2012 Nov;60(5):1148-56. doi: 10.1161/HYPERTENSIONAHA.112.196980. Epub 2012 Sep 24. PMID 23006736
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262